CLINICAL TRIAL: NCT06780306
Title: A Phase 2 Randomized, Controlled, Multicenter, Dose Optimization Study of TTAX03 in the Treatment of Mild to Moderate Dry Eye Disease (DED)
Brief Title: A Study in the Treatment of Mild to Moderate Dry Eye Disease Comparing Saline to TTAX03.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTAX03-CR010
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye; Dry Eye Disease (DED); Dry Eye Disease With Severe Keratitis
Keywords: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10mg TTAX03 reconstituted in 150 uL saline (Experimental): For all four groups, 100 mL of reconstituted solution will be applied into the concave bowl of a bandage contact lens and inserted into the study eye.
  Interventions: Biological: TTAX03
- 10mg TTAX03 reconstituted in 300 uL saline (Active Comparator): For all four groups, 100 mL of reconstituted solution will be applied into the concave bowl of a bandage contact lens and inserted into the study eye.
  Interventions: Biological: TTAX03
- 10mg TTAX03 reconstituted in 600 uL saline (Active Comparator): For all four groups, 100 mL of reconstituted solution will be applied into the concave bowl of a bandage contact lens and inserted into the study eye.
  Interventions: Biological: TTAX03
- 300 uL of saline (Placebo Comparator): For all four groups, 100 mL of reconstituted solution will be applied into the concave bowl of a bandage contact lens and inserted into the study eye.
  Interventions: Biological: Saline (NaCl 0,9 %) (placebo)

INTERVENTIONS:
Biological: TTAX03 — Lyophilized and Micronized Particulate Human Amniotic and Umbilical Cord
  Arms: 10mg TTAX03 reconstituted in 150 uL saline; 10mg TTAX03 reconstituted in 300 uL saline; 10mg TTAX03 reconstituted in 600 uL saline
Biological: Saline (NaCl 0,9 %) (placebo) — 300 mL Sterile, preservative free 0.9% NaCl
  Arms: 300 uL of saline

SUMMARY:
The purpose of this randomized, controlled, multicenter study is to evaluate the safety and efficacy of TTAX03 in participants with mild to moderate DED.

The primary question it aims to answer is if TTAX03 is safe. The secondary is the effectiveness.

Researchers will compare 10mg of TTAX03 reconstituted in 150, 300, or 600 uL saline to the saline control group to look at effectiveness.

Participants will be randomized to a treatment group one time and be evaluated at 5 different study visits.

DETAILED DESCRIPTION:
The purpose of this randomized, controlled, multicenter study is to evaluate the safety and efficacy of TTAX03 in participants with mild to moderate DED. After confirmation of inclusion and exclusion criteria, all eligible patients will be randomized in a 1:1:1:1 ratio to receive one of the three doses of TTAX03 (10 mg of TTAX03 reconstituted in 150, 300, or 600 uL saline, i.e., subgroup A, B, and C, respectively) or to the saline control group (subgroup D). For all four groups, the same volume of reconstituted solution will be applied into the concave bowl of a bandage contact lens and inserted into the eye. The more severe eye will serve as the study eye, which meets inclusion and exclusion criteria. The treatment period is 5 days of continuous bandage contact lens wear. Safety follow-up without further treatment will continue for twelve weeks. After baseline (day 1) and completion of treatment, enrolled patients will be evaluated for safety and efficacy at Day 6 ± 1, Day 29 ± 3, Day 57 ± 3, and Day 85 ± 3.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Provision of signed and dated informed consent form.
3. Baseline VAS Dryness score ≥40
4. Baseline Ocular Surface Disease Index (OSDI) score ≥ 13.
5. Baseline corneal fluorescein staining with a total score ≥ 4 but ≤13, and ≥ 2 in at least one region, by the NEI Grading System† in the study eye.
6. In the opinion of the investigator, the participant can follow oral and written instructions.
7. In the opinion of the investigator, the participant can complete all study procedures and visits.

Exclusion Criteria:

1. Has a corneal ectatic disorder or other ocular surface disease such as limbal stem cell deficiency or a cicatricial component (e.g., symblepharon, fornix foreshortening and lid margin/lashes abnormality) caused for example by oGVHD, irradiation, chemical burns, trachoma, Stevens Johnson syndrome/toxic epidermal necrolysis, ocular cicatricial pemphigoid, or the destruction of conjunctival goblet cells (as with vitamin A deficiency).
2. Has severe blepharitis or severe obvious inflammation of the lid margin.
3. Has severe conjunctivochalasis.
4. Has nocturnal exposure e.g. incomplete closure or lagophthalmos or floppy eyelid.
5. Has epithelial basement membrane dystrophy (i.e., map-dot-fingerprint dystrophy) or history of recurrent corneal erosion
6. Has neuropathic corneal pain
7. Has a sunken globe (due to the reduction or loss of orbital fat)
8. Has severe DED per corneal fluorescein staining with a total score ≥ 13by the NEI Grading System in either eye.
9. Prior history of intolerance or adverse events using BCL.
10. Have had dissolvable or temporary plug(s) (including hydrogel or Lacrifill®) inserted within 6 months prior to screening.
11. Is using a nasal cholinergic agonist such as Tyrvaya in the last 30 days.
12. Has had previous ocular surgery in the study eye within the past 12 weeks.
13. Plans to use autologous serum drops during the study period in either eye.
14. Has elevated intraocular pressure >21mmHg in either eye requiring topical therapy.
15. Is currently using or plans to use topical glaucoma medication in either eye.
16. Has a known allergy to topical ophthalmic sodium fluorescein dye.
17. Has a known intolerance to unbuffered normal saline.
18. Prior adverse events of using human birth tissue product.
19. Is currently incarcerated or anticipates possible incarceration during the time course of this study.
20. Has tested positive for COVID-19 within 28 days prior to screening.
21. Is currently participating in any other type of eye-related clinical or research study that in the opinion of the investigator would confound or would risk confounding study results.
22. Has a condition or is in a situation which, in the investigator's opinion, may put the participant at significant risk, may confound study outcomes, or may significantly interfere with the participant's participation in the study.
23. Prior amniotic membrane product used for dry eye therapy in the study eye in the past 6 months.
24. Has Strabismus (squint/crossed eyes) or Amblyopia (lazy eye).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Determine 12 week ocular and general safety after application of TTAX03. | 12 weeks
  Incidence and nature of treatment emergent adverse events (TEAE) between TTAX03 and saline.

SECONDARY OUTCOMES:
Proportion of participants who show complete resolution of superficial punctate keratopathy, i.e., absence of corneal fluorescein staining, on Day 6 by group. | Day 6
  Determine the relationship between TTAX03 doses and efficacy per changes from baseline in complete resolution of superficial punctate keratopathy (defined by corneal fluorescein staining) at Day 6 when compared to the saline control.
Mean change from baseline to Day 6 in corneal fluorescein staining (National Eye Institute (NEI) score) by group. | Baseline to Day 6
  Examine the relationship between TTAX03 doses and changes from baseline in corneal epithelial staining at Day 6 when compared to the saline control.
Proportion of participants with clinically meaningful reduction in corneal fluorescein staining (NEI ≥ 3) from baseline to Day 6 by group. | Baseline to Day 6
  Examine the relationship between TTAX03 doses and clinically meaningful changes from baseline vs. saline in corneal staining during the follow up to 12 weeks.
Proportion of participants with clinically meaningful reduction in corneal fluorescein staining (NEI ≥ 3) from baseline to Day 29 by group. | Baseline to Day 29
  Examine the relationship between TTAX03 doses and clinically meaningful changes from baseline vs. saline in corneal staining during the follow up to 12 weeks.
Proportion of participants with clinically meaningful reduction in corneal fluorescein staining (NEI ≥ 3) from baseline to Day 57 by group. | Baseline to Day 57
  Examine the relationship between TTAX03 doses and clinically meaningful changes from baseline vs. saline in corneal staining during the follow up to 12 weeks.
Proportion of participants with clinically meaningful reduction in corneal fluorescein staining (NEI ≥ 3) from baseline to Day 85 by group. | Baseline to Day 85
  Examine the relationship between TTAX03 doses and clinically meaningful changes from baseline vs. saline in corneal staining during the follow up to 12 weeks.
Mean change in dry eye symptoms (measured by OSDI) from baseline on Day 6 by group. | Baseline to Day 6
  Examine the relationship between TTAX03 doses and change of dry eye symptoms from baseline when compared to saline at Day 6.
Mean change in dry eye symptoms (measured by VAS) from baseline on Day 6 by group. | Baseline to Day 6
  Examine the relationship between TTAX03 doses and change of dry eye symptoms from baseline when compared to saline at Day 6.
Mean change from baseline in BCVA (logMAR) measured by ETDRS chart on Day 6 by group. | Baseline to Day 6
  Examine the relationship between TTAX03 doses and change of best corrected visual acuity (BCVA) from baseline when compared to saline at Day 6.
Proportion of participants who show complete resolution of superficial punctate keratopathy, i.e., absence of corneal fluorescein staining, on Day 29 by group. | Day 29
  Examine the relationship between TTAX03 doses and percentages of participants showing complete resolution of corneal staining from baseline when compared to saline during the follow up 12 weeks.
Proportion of participants who show complete resolution of superficial punctate keratopathy, i.e., absence of corneal fluorescein staining, on Day 57 by group. | Day 57
  Examine the relationship between TTAX03 doses and percentages of participants showing complete resolution of corneal staining from baseline when compared to saline during the follow up 12 weeks.
Proportion of participants who show complete resolution of superficial punctate keratopathy, i.e., absence of corneal fluorescein staining, on Day 85 by group. | Day 85
  Examine the relationship between TTAX03 doses and percentages of participants showing complete resolution of corneal staining from baseline when compared to saline during the follow up 12 weeks.
Mean change from baseline in corneal fluorescein staining (National Eye Institute (NEI) score) on Day 29 by group. | Baseline to Day 29
  Examine the relationship between TTAX03 doses and change of corneal epithelial staining from baseline between when compared to saline during the follow up to 12 weeks.
Mean change from baseline in corneal fluorescein staining (National Eye Institute (NEI) score) on Day 57 by group. | Baseline to Baseline to Day 57
  Examine the relationship between TTAX03 doses and change of corneal epithelial staining from baseline between when compared to saline during the follow up to 12 weeks.
Mean change from baseline in corneal fluorescein staining (National Eye Institute (NEI) score) on Day 85 by group. | Baseline to Baseline to Day 85
  Examine the relationship between TTAX03 doses and change of corneal epithelial staining from baseline between when compared to saline during the follow up to 12 weeks.
Mean change in dry eye symptoms (measured by OSDI) from baseline on Day 29 by group. | Baseline to Day 29
  Examine the relationship between TTAX03 doses and change of ocular dry eye symptoms from baseline when compared to saline during the follow up to 12 weeks.
Mean change in dry eye symptoms (measured by OSDI) from baseline on Day 57 by group. | Baseline to Day 57
  Examine the relationship between TTAX03 doses and change of ocular dry eye symptoms from baseline when compared to saline during the follow up to 12 weeks.
Mean change in dry eye symptoms (measured by OSDI) from baseline on Day 85 by group. | Baseline to Day 85
  Examine the relationship between TTAX03 doses and change of ocular dry eye symptoms from baseline when compared to saline during the follow up to 12 weeks.
Mean change in dry eye symptoms (measured by VAS) from baseline on Day 29 by group. | Baseline to Day 29
  Examine the relationship between TTAX03 doses and change of ocular dry eye symptoms from baseline when compared to saline during the follow up to 12 weeks.
Mean change in dry eye symptoms (measured by VAS) from baseline on Day 57 by group. | Baseline to Day 57
  Examine the relationship between TTAX03 doses and change of ocular dry eye symptoms from baseline when compared to saline during the follow up to 12 weeks.
Mean change in dry eye symptoms (measured by VAS) from baseline on Day 85 by group. | Baseline to Day 85
  Examine the relationship between TTAX03 doses and change of ocular dry eye symptoms from baseline when compared to saline during the follow up to 12 weeks.
Mean change from baseline in BCVA (logMAR) measured by ETDRS chart on Days 29 by group. | Day 29
  Examine the relationship between TTAX03 doses and change of BCVA from baseline when compared to saline during the follow up to 12 weeks.
Mean change from baseline in BCVA (logMAR) measured by ETDRS chart on Day 57 by group. | Day 57
  Examine the relationship between TTAX03 doses and change of BCVA from baseline when compared to saline during the follow up to 12 weeks.
Mean change from baseline in BCVA (logMAR) measured by ETDRS chart on Day 85 by group. | Day 85
  Examine the relationship between TTAX03 doses and change of BCVA from baseline when compared to saline during the follow up to 12 weeks.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University California Berkeley, Berkeley, California
  - Advanced Research, LLC., Deerfield Beach, Florida
  - Southwest Eye Care, Chaska, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Eye Associates of North Jersey, Dover, New Jersey
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - Wilmington Eye at Brunswick Forest, Leland, North Carolina
  - CORE, Inc. / Vita Eye Clinic, Shelby, North Carolina
  - Westlake Eye Specialists, Austin, Texas